CLINICAL TRIAL: NCT05837988
Title: Construction of Symptom Network in Maintenance Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-071-B
Record Dates: First submitted 2023-04-17; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Symptom Cluster; Symptoms and Signs; Hemodialysis Complication; Hemodialysis-Associated Pruritus
Keywords: Symptom Network; Hemodialysis; Symptom Burden; Symptom Management
MeSH Terms: conditions — Syndrome; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MHD patients: Cross sectional survey, no intervention measures involved

SUMMARY:
Through a cross-sectional questionnaire survey, a general information questionnaire and Dialysis Frequency, Severity, and Symptom Burden Index were used to investigate the frequency, severity, and degree of symptom distress in MHD patients, and to analyze the differences in symptom distress status between long and short dialysis age MHD patients. Using the R 4.2.2 software qgraph package, construct symptom networks for MHD patients of long and short dialysis age through network analysis. Analyze network centrality indicators, including intensity, closeness centrality, and mediation centrality, to identify core symptoms and compare if there are any differences between the two groups, aiming to lay the foundation for precise and efficient phased symptom management.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) is caused by various kidney diseases, leading to irreversible decline in renal function. The main renal replacement therapy (RRT) for ESRD is hemodialysis (HD), peritoneal dialysis (PD), and kidney transplantation. Due to the impact of kidney supply on kidney transplantation, it is limited in clinical practice, and hemodialysis has become the most common method of RRT in most countries. According to the registration system of the Chinese Research Data Services (CNRDS), as of the end of 2021, there were 751098 dialysis patients and 155738 new patients in China, with an average dialysis age of 50.9 months. The proportion of patients with dialysis age greater than 5 years was 31.5%. There are a large number of hemodialysis patients with a longer dialysis age.

With the continuous development of dialysis technology, the survival rate of maintenance hemodialysis (MHD) patients is becoming higher and higher. However, MHD patients may experience various symptoms during long-term treatment, which is the main cause of discomfort and physical and mental health for patients. The physical and mental pain or torment experienced by patients due to the disease itself and/or the symptoms caused by treatment is called symptom distress. Multiple studies have shown that the incidence of symptom distress in MHD patients ranges from 13.75% to 91.5%, which is at a high level. Symptom distress is negatively correlated with the quality of life of MHD patients. Excessive symptom distress increases the cost of treatment and exacerbates the psychological burden on patients. Persistent symptom burden can significantly affect the quality of life of MHD patients and increase their mortality rate. MHD patients suffer from multiple symptoms at the same time. Li Jiuhong et al.'s research results show that MHD patients experience a total of 3-25 (13.12 ± 5.27) symptoms, which is similar to Weisbord et al.'s average of 9 symptoms. MHD patients experience a wide variety of symptoms, and how to accurately and effectively manage symptoms is the future research direction.

With the prolongation of dialysis treatment time for patients, some urea toxin that cannot be completely cleared by dialysis accumulates in the patient's body, which is closely related to discomfort symptoms such as itching, joint pain, and difficulty falling asleep. Ran Yuli et al. found that the dialysis age of MHD patients is negatively correlated with their physical function and role. With the prolongation of dialysis age, the physiological function of MHD patients will decrease to varying degrees, and various disease-related complications will also occur. The focus of symptom management will shift accordingly. Conducting grouping studies based on dialysis age for MHD patients has certain clinical significance. At present, domestic scholars use a 5-year hemodialysis period as the boundary, dividing dialysis age>5 years into long dialysis age, and dialysis age ≤ 5 years into short dialysis age. Hu Qian and others set up symptom management consultants to develop symptom management pathways and guide responsible nurses to implement symptom management for patients according to the pathway table. The results indicate that setting up symptom management consultants can reduce the incidence of symptoms in MHD patients, improve their quality of life, and improve patient satisfaction. A meta-analysis showed that aerobic exercise can improve several symptoms related to hemodialysis in adults receiving MHD, including restless leg syndrome, depressive symptoms, muscle spasms, and fatigue. Zhao Ying et al. used air wave pressure therapy to prevent dialysis related muscle spasms, Zuo et al. managed symptoms of fatigue through nurse led non drug multidisciplinary holistic care, Beerappa et al. improved sleep disorders in MHD patients through aromatherapy, Guo Junjun et al. improved fatigue symptoms and alleviated sleep disorders in MHD patients through acupoint massage. When conducting symptom management for MHD patients, existing studies have not distinguished the age of dialysis, and currently, symptom management for MHD patients mainly focuses on a single symptom or symptom group, ignoring the interaction between multiple symptoms in the real world. In real clinical situations, patients often have multiple symptoms at the same time, and it is urgent to identify the core symptoms of patients to improve the accuracy and efficiency of symptom management.

With the development of information technology, big data analysis technology, and the innovation of complex scientific research concepts in the real world, the concept of symptom networks is gradually replacing the previous research paradigm that focuses on individual symptoms and must control other variables. Symptom network is a collective representation of symptoms related to a patient's disease, and based on complex network analysis to quantitatively study the correlation between different symptoms. It studies the network structure, nodes, and network indicators composed of individual symptoms to reflect the interaction mechanism of symptoms in the real world and provide precise intervention targets. Discovering core symptom targets through symptom networks can improve the management efficiency and intervention accuracy of symptom management, evolving from the working mode of "having multiple symptoms and providing multiple sets of intervention measures" to "identifying intervention targets and providing intervention measures targeting target symptoms". Since Fried et al. first proposed the concept of symptom networks in 2015, the research paradigm of symptom networks has been applied in psychopathology, chronic disease symptom management, long-term follow-up of tumors, and patient self-management. Lin et al. constructed a self-reported psychological and neurological symptom network for head and neck cancer patients through network analysis. The results showed that network analysis clarified the interrelationships between five psychological and neurological symptoms, and identified depression as the core symptom. It is recommended to develop symptom management measures for depression in clinical practice. Han et al. constructed symptom networks for autism and schizophrenia. Yang Hongli et al. applied symptom networks to HIV infected individuals and identified fatigue as the core symptom. They suggested that when HIV infected individuals have multiple symptoms at the same time, high-intensity and precise intervention on fatigue can reduce the transmission of fatigue as a mediating bridge in the symptom network, reduce the severity of fatigue symptoms, and also alleviate the severity of other symptoms. As mentioned above, symptom network analysis can identify core symptoms, and changing these core symptoms may be an important entry point for changing the entire network. In practical clinical work, implementing key interventions by nurses on core symptoms can more effectively improve other related symptoms and improve intervention efficiency. Applying symptom networks to the field of symptom management is a promising and precise technology in real-world clinical settings.

This study has developed a symptom distress questionnaire for maintenance hemodialysis patients. Previous literature on symptom distress and symptom management in MHD patients has been reviewed. Whether there are differences in symptom distress among MHD patients of different dialysis ages, and how to identify the core symptoms of MHD patients of different dialysis ages through symptom networks to improve the accuracy and effectiveness of intervention are all directions that need to be studied in the future. The research hypotheses of this study are: ① There are differences in the frequency, severity, and degree of symptom distress between long and short dialysis age MHD patients; ② By using network analysis methods to construct symptom networks for long and short dialysis age MHD patients, identify the core symptoms of different dialysis age MHD patients. Based on literature review and clinical experience, it is assumed that the core symptoms of long dialysis age MHD patients are itching or dry skin, while the core symptoms of short dialysis age MHD patients are fatigue or dry mouth.

ELIGIBILITY:
Inclusion Criteria:

* Age not less than 18 years old;
* Regular hemodialysis time greater than or equal to 3 months;
* The dialysis plan did not change within one month;
* Informed consent and voluntary participation in this study.

Exclusion Criteria:

* Previous or current mental illness;
* Cognitive impairment;
* Acute cardiovascular and cerebrovascular disease;
* Acute infection period;
* Complications such as severe cerebrovascular sequelae and tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are maintenance hemodialysis patients selected by convenience sampling method from six blood purification centers, including the East, West, South, Baoshan Branch of Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Ningbo Hangzhou Bay Hospital, and Punan Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Estimated)
Dates: Start 2023-05-08 (Estimated); Primary Completion 2023-05-08 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
symptom burden | at the time of patient enrollment
  Through a cross-sectional questionnaire survey, the Dialysis Frequency, Severity, and Symptom Burden Index were used to investigate the frequency, severity, and degree of symptom distress in MHD patients, and to analyze the differences in symptom distress status between long and short dialysis age MHD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tingting Liu, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Result] Pippias M, Stel VS, Abad Diez JM, Afentakis N, Herrero-Calvo JA, Arias M, Tomilina N, Bouzas Caamano E, Buturovic-Ponikvar J, Cala S, Caskey FJ, Castro de la Nuez P, Cernevskis H, Collart F, Alonso de la Torre R, Garcia Bazaga Mde L, De Meester J, Diaz JM, Djukanovic L, Ferrer Alamar M, Finne P, Garneata L, Golan E, Gonzalez Fernandez R, Gutierrez Avila G, Heaf J, Hoitsma A, Kantaria N, Kolesnyk M, Kramar R, Kramer A, Lassalle M, Leivestad T, Lopot F, Macario F, Magaz A, Martin-Escobar E, Metcalfe W, Noordzij M, Palsson R, Pechter U, Prutz KG, Ratkovic M, Resic H, Rutkowski B, Santiuste de Pablos C, Spustova V, Suleymanlar G, Van Stralen K, Thereska N, Wanner C, Jager KJ. Renal replacement therapy in Europe: a summary of the 2012 ERA-EDTA Registry Annual Report. Clin Kidney J. 2015 Jun;8(3):248-61. doi: 10.1093/ckj/sfv014. Epub 2015 Mar 23. PMID 26034584
- [Result] Thurlow JS, Joshi M, Yan G, Norris KC, Agodoa LY, Yuan CM, Nee R. Global Epidemiology of End-Stage Kidney Disease and Disparities in Kidney Replacement Therapy. Am J Nephrol. 2021;52(2):98-107. doi: 10.1159/000514550. Epub 2021 Mar 22. PMID 33752206
- [Result] McCorkle R, Young K. Development of a symptom distress scale. Cancer Nurs. 1978 Oct;1(5):373-8. No abstract available. PMID 250445
- [Result] You AS, Kalantar SS, Norris KC, Peralta RA, Narasaki Y, Fischman R, Fischman M, Semerjian A, Nakata T, Azadbadi Z, Nguyen DV, Kalantar-Zadeh K, Rhee CM. Dialysis symptom index burden and symptom clusters in a prospective cohort of dialysis patients. J Nephrol. 2022 Jun;35(5):1427-1436. doi: 10.1007/s40620-022-01313-0. Epub 2022 Apr 16. PMID 35429297
- [Result] Wang X, Shi Q, Mo Y, Liu J, Yuan Y. Palliative care needs and symptom burden in younger and older patients with end-stage renal disease undergoing maintenance hemodialysis: A cross-sectional study. Int J Nurs Sci. 2022 Oct 4;9(4):422-429. doi: 10.1016/j.ijnss.2022.09.015. eCollection 2022 Oct. PMID 36285085
- [Result] Weisbord SD, Fried LF, Arnold RM, Fine MJ, Levenson DJ, Peterson RA, Switzer GE. Prevalence, severity, and importance of physical and emotional symptoms in chronic hemodialysis patients. J Am Soc Nephrol. 2005 Aug;16(8):2487-94. doi: 10.1681/ASN.2005020157. Epub 2005 Jun 23. PMID 15975996
- [Result] Hargrove N, El Tobgy N, Zhou O, Pinder M, Plant B, Askin N, Bieber L, Collister D, Whitlock R, Tangri N, Bohm C. Effect of Aerobic Exercise on Dialysis-Related Symptoms in Individuals Undergoing Maintenance Hemodialysis: A Systematic Review and Meta-Analysis of Clinical Trials. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):560-574. doi: 10.2215/CJN.15080920. Epub 2021 Mar 25. PMID 33766925
- [Result] Zuo M, Zhu W, Lin J, Zhuo J, He X, Jing X, Tang J, Deng R. The impact of nurse-led nonpharmacological multidisciplinary holistic nursing care on fatigue patients receiving hemodialysis: a randomized, parallel-group, controlled trial. BMC Nurs. 2022 Dec 12;21(1):352. doi: 10.1186/s12912-022-01126-3. PMID 36503477
- [Result] Beerappa H, Gt K, Chandrababu R. The Effects of Inhalational Lavender Essential Oil Aromatherapy on Sleep Quality in Hemodialysis Patients: A Before-and-After-Intervention Trial. Holist Nurs Pract. 2023 Nov-Dec 01;37(6):356-362. doi: 10.1097/HNP.0000000000000521. Epub 2022 Jun 1. PMID 35703289
- [Result] Fried EI, Boschloo L, van Borkulo CD, Schoevers RA, Romeijn JW, Wichers M, de Jonge P, Nesse RM, Tuerlinckx F, Borsboom D. Commentary: "Consistent Superiority of Selective Serotonin Reuptake Inhibitors Over Placebo in Reducing Depressed Mood in Patients with Major Depression". Front Psychiatry. 2015 Aug 21;6:117. doi: 10.3389/fpsyt.2015.00117. eCollection 2015. No abstract available. PMID 26347663
- [Result] Kachadourian LK, Harpaz-Rotem I, Tsai J, Southwick SM, Pietrzak RH. Posttraumatic Stress Disorder Symptoms, Functioning, and Suicidal Ideation in US Military Veterans: A Symptomics Approach. Prim Care Companion CNS Disord. 2019 Apr 25;21(2):18m02402. doi: 10.4088/PCC.18m02402. PMID 31050228
- [Result] Lin Y, Bruner DW, Paul S, Miller AH, Saba NF, Higgins KA, Shin DM, Zhang W, Miaskowski C, Xiao C. A network analysis of self-reported psychoneurological symptoms in patients with head and neck cancer undergoing intensity-modulated radiotherapy. Cancer. 2022 Oct;128(20):3734-3743. doi: 10.1002/cncr.34424. Epub 2022 Aug 15. PMID 35969226
- [Result] Han GT, Trevisan DA, Foss-Feig J, Srihari V, McPartland JC. Distinct Symptom Network Structure and Shared Central Social Communication Symptomatology in Autism and Schizophrenia: A Bayesian Network Analysis. J Autism Dev Disord. 2023 Sep;53(9):3636-3647. doi: 10.1007/s10803-022-05620-0. Epub 2022 Jun 25. PMID 35752729
- [Result] Danquah FV, Zimmerman L, Diamond PM, Meininger J, Bergstrom N. Frequency, severity, and distress of dialysis-related symptoms reported by patients on hemodialysis. Nephrol Nurs J. 2010 Nov-Dec;37(6):627-38; quiz 639. PMID 21290917
- [Result] Dodd MJ, Miaskowski C, Paul SM. Symptom clusters and their effect on the functional status of patients with cancer. Oncol Nurs Forum. 2001 Apr;28(3):465-70. PMID 11338755
- [Result] Weisbord SD, Fried LF, Arnold RM, Rotondi AJ, Fine MJ, Levenson DJ, Switzer GE. Development of a symptom assessment instrument for chronic hemodialysis patients: the Dialysis Symptom Index. J Pain Symptom Manage. 2004 Mar;27(3):226-40. doi: 10.1016/j.jpainsymman.2003.07.004. PMID 15010101
- [Result] Papachristou N, Barnaghi P, Cooper B, Kober KM, Maguire R, Paul SM, Hammer M, Wright F, Armes J, Furlong EP, McCann L, Conley YP, Patiraki E, Katsaragakis S, Levine JD, Miaskowski C. Network Analysis of the Multidimensional Symptom Experience of Oncology. Sci Rep. 2019 Feb 19;9(1):2258. doi: 10.1038/s41598-018-36973-1. PMID 30783135
- [Result] Dicenso A, Bayley L, Haynes RB. Accessing pre-appraised evidence: fine-tuning the 5S model into a 6S model. Evid Based Nurs. 2009 Oct;12(4):99-101. doi: 10.1136/ebn.12.4.99-b. No abstract available. PMID 19779069
- [Result] Brouwers MC, Kho ME, Browman GP, Burgers JS, Cluzeau F, Feder G, Fervers B, Graham ID, Grimshaw J, Hanna SE, Littlejohns P, Makarski J, Zitzelsberger L; AGREE Next Steps Consortium. AGREE II: advancing guideline development, reporting and evaluation in health care. CMAJ. 2010 Dec 14;182(18):E839-42. doi: 10.1503/cmaj.090449. Epub 2010 Jul 5. No abstract available. PMID 20603348
- [Result] Pearson A, Wiechula R, Court A, Lockwood C. The JBI model of evidence-based healthcare. Int J Evid Based Healthc. 2005 Sep;3(8):207-15. doi: 10.1111/j.1479-6988.2005.00026.x. PMID 21631749
- [Result] van Borkulo CD, Borsboom D, Epskamp S, Blanken TF, Boschloo L, Schoevers RA, Waldorp LJ. A new method for constructing networks from binary data. Sci Rep. 2014 Aug 1;4:5918. doi: 10.1038/srep05918. PMID 25082149
- [Result] Altenbuchinger M, Weihs A, Quackenbush J, Grabe HJ, Zacharias HU. Gaussian and Mixed Graphical Models as (multi-)omics data analysis tools. Biochim Biophys Acta Gene Regul Mech. 2020 Jun;1863(6):194418. doi: 10.1016/j.bbagrm.2019.194418. Epub 2019 Oct 19. PMID 31639475

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT05837988/Prot_SAP_000.pdf